CLINICAL TRIAL: NCT02800044
Title: Studying the Effectiveness of Non-Invasive Glucose Sensors in Patients With Diabetes: The SENSOR Study
Acronym: SENSOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results were not accurate; despite multiple efforts to troubleshoot.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward Chao, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: UCSDSOM
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing glucose sensor (Experimental): The study team will measure glucose readings from the non-invasive sensor and from a glucometer at the following time points: fasting, 1.5 to 2 hours after a meal, and before and after 15-30 minutes of pedaling on a stationary bicycle at 80% maximum heart rate..
  Interventions: Device: Wearing a non-invasive glucose sensor

INTERVENTIONS:
Device: Wearing a non-invasive glucose sensor — Glucose readings will be obtained from both a glucometer (fingerstick readings) and from the non-invasive glucose sensor at the following four timepoints: fasting, 1.5 to 2 hours after consuming a meal, and before and after 15-30 minutes of moderate exercise on a stationary bicycle.

SUMMARY:
The overall goal for this pilot clinical trial is to explore the accuracy and acceptability of a non-invasive, wearable glucose sensor in patients living with DM. This study will compare needleless glucose sensor readings with glucometer measurements from patients with type 1 or type 2 diabetes (T1DM or T2DM), under varying conditions.

DETAILED DESCRIPTION:
Self-monitoring of blood glucose (SMBG) can both facilitate and hinder adherence in patients with diabetes mellitus (DM). Readings provide real-time information on hypoglycemic and hyperglycemic excursions. These data are crucial to successfully managing this disease, as SMBG can help guide decisions on titrating medications, and can potentially encourage patient engagement. There are drawbacks. Piercing the skin to check glucose up to several times a day can be uncomfortable and obtrusive for a patient with DM. SMBG offers only a snapshot of the patient's glucose at the time of testing.

Continuous glucose monitoring (CGM) can reveal glucose trends. A subcutaneous sensor transmits interstitial glucose readings approximately every five minutes. Yet, sensor insertion requires a needle. Patients still must test SMBG about 4 times per day to calibrate the CGM sensor. This modality is less accurate with low or rapidly rising glucose. CGM is also not widely available, due to cost and insurance issues. A non-invasive glucose monitor, the GlucoWatch, was discontinued due to problems with accuracy and tolerability.

Compounding these challenges is the surging number of individuals with DM. Every 19 seconds, an American 20 years of age or older is diagnosed with DM. If current trends continue, 1 in 3 Americans could have DM by 2050.

There is thus an unmet need for a non-invasive glucose monitoring device. UCSD nanoengineers developed a flexible, ultra-thin sensor adherent to the skin, similar to a temporary tattoo. Preliminary data from seven individuals without DM demonstrated correlation between glucose measurements from this sensor and a glucometer. Evaluating this sensor in patients with DM will be critical: while hour-to-hour blood glucose fluctuates approximately 50% throughout the day in those without DM, it may vary up to 10-fold in patients with DM. This study would be the first to examine this sensor in individuals with DM. The investigators hypothesize that compared with a glucometer, a tattoo sensor can accurately measure glucose in patients with DM.

ELIGIBILITY:
Inclusion Criteria:

1. An existing diagnosis of diabetes mellitus, either T1DM or T2DM
2. Absence of cognitive impairment, as demonstrated by a Montreal Cognitive Assessment (MOCA) score greater than 26; those individuals with questionable cognitive ability will be screened with this instrument.
3. Ability to provide informed consent for participation.

Exclusion Criteria:

1. Individuals without diabetes
2. Those who have a MOCA score of 26 or less
3. Those who cannot speak or read English. The investigators are limiting participation to those who read and speak English, as this is a pilot study of a small number of participants, that will very unlikely offer the prospect of direct benefit from participating.
4. Individuals who have a cardiac, respiratory, or other condition that would preclude safely exercising at a moderate pace. Along with a medical history and physical examination by the PI, prospective participants will complete the Physical Activity Readiness Questionnaire (PAR-Q) to help determine those who may safely exercise for this study. One or more "yes" responses does not necessarily exclude an individual from participating.
5. Individuals who have frequent hypoglycemia, hypoglycemia unawareness, or who are at high risk for hypoglycemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
accuracy | 1 year
  how the non-invasive glucose sensor measurements correlate with glucometer readings

SECONDARY OUTCOMES:
acceptability | 1 year
  how acceptable patients find this sensor

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Chao, DO, Principal Investigator — UCSD
Locations (1):
- UCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandodkar AJ, Jia W, Yardimci C, Wang X, Ramirez J, Wang J. Tattoo-based noninvasive glucose monitoring: a proof-of-concept study. Anal Chem. 2015 Jan 6;87(1):394-8. doi: 10.1021/ac504300n. Epub 2014 Dec 12. PMID 25496376

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT02800044/Prot_SAP_000.pdf